CLINICAL TRIAL: NCT05916092
Title: A Prospective, Multicenter, Post Market Surveillance Study on a Modular SI Joint Fusion System
Brief Title: Post-Market Clinical Study on a Modular SI Joint Fusion System
Acronym: SPARTAN
Status: Enrolling by invitation | Type: Observational
Sponsor: CornerLoc (Industry)
Responsible Party: Sponsor
Other Study IDs: SPARTAN-001
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Sacroiliitis; Sacroiliac Joint Dysfunction
MeSH Terms: conditions — Sacroiliitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Lateral-Oblique TransLoc 3D Screw(s): Patients receiving the TransLoc 3D Screw(s) version will receive screw(s) placed lateral-obliquely into the intended SI joint.
  Interventions: Device: TransLoc 3D
- Lateral Oblique TransLoc 3D Screw with Posterior Device (Hybrid): Patients receiving the TransLoc 3D Hybrid construct will receive one 3D-printed titanium screw placed lateral-obliquely and one 3D-printed titanium posterior device across the same sacroiliac joint.
  Interventions: Device: TransLoc 3D

INTERVENTIONS:
Device: TransLoc 3D — TransLoc 3D SI Joint Fusion System

SUMMARY:
A prospective study on the use of the TransLoc 3D SI Joint Fusion System for patients with sacroiliac joint disruptions or degenerative sacroiliitis.

DETAILED DESCRIPTION:
Multicenter, prospective, post-market surveillance study on the TransLoc 3D Sacroiliac Joint Fusion System including two treatment arms: 1) Lateral-Oblique TransLoc 3D Screw(s), 2) Lateral Oblique TransLoc 3D Screw with Posterior Device (Hybrid). Data from this post-market study will be used to support knowledge of clinical efficacy and improvement with the use of TransLoc 3D Sacroiliac Joint Fusion System.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following inclusion criteria by the end of the screening phase should be considered for admission to the study:

  * Age 18-85* (*Over 85 is allowed with H&P assessment screening upon approval by Medical Monitor);
  * Absent condition of high-risk surgical candidate (see training manual for definition);
  * Patient has lower back pain with a confirmed diagnosis of sacroiliac joint disruption or degenerative sacroiliitis for a period of >6 months and who has not responded to optimal conservative care (PT or prescribed HEP, optimal medical management including NSAIDs);
  * Diagnosis of sacroiliac joint disruption or degenerative sacroiliitis based on ALL of the following: a. Patient has pain at or close to the posterior superior iliac spine (PSIS) with possible radiation into buttocks, posterior thigh or groin and can point with a single finger to the location of pain (Fortin Finger Test), and b. at least three positive findings with provocative maneuvers (FABER, Gaenslen, Thigh Thrust or Posterior Shear, SI Compression, SI Distraction, and Yeoman Test);
  * Patient has a diagnostic SIJ injection (SIJI) that provided a minimum of 75% relief of primary (index) pain with the diagnostic SIJI on two separate occasions;
  * Patient meets Medicare and payer requirements for medical necessity, see detailed requirements in training manual;
  * SI joint disruption: Asymmetric SI joint widening on X-ray or CT scan or degenerative sacroiliitis with radiographic evidence of SIJ degeneration as evidenced on CT or X-ray;
  * SI joint pain or instability with or without prior lumbar/lumbosacral surgery;
  * Baseline Oswestry Disability Index (ODI) score of at least 30%;
  * Baseline SI joint pain score of at least 60 on 0-100mm visual analog scale (or at least a 6 on NRS);
  * Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements;
  * Failed SIJ fusion revisions can be included if all other inclusion criteria are met;
  * Patient must be able to communicate with study personnel via phone, text, or email;
  * PI must confirm women of childbearing years are not pregnant or plan to become pregnant prior to surgery;
  * Cardiac Clearance for patients with diagnosis of cardiac disease;
  * Patient has signed study-specific informed consent form.

Exclusion Criteria:

* Patient will not be entered into the study if they meet one of the following criteria:

  * Current severe back pain due to other causes, such as lumbar disc degeneration, lumbar disc herniation, lumbar spondylolisthesis, lumbar spinal stenosis, lumbar facet degeneration, lumbar radicular pain that extends beyond the mid-thigh, and lumbar vertebral body fracture;
  * SIJ pain secondary to inflammatory conditions or other known sacroiliac pathology such as: Sacral dysplasia, Inflammatory sacroiliitis (e.g., ankylosing spondylitis or other HLA-associated spondylo-arthropathy), Tumor or infection in the SI joint, Acute fracture or Crystal arthropathy;
  * History of recent (<1 year) major trauma to pelvis (MVA or significant accident that results in acute injury to pelvis requiring hospitalization or surgery);
  * Previously diagnosed osteoporosis (defined as prior T-score <-2.5 or history of osteoporotic fracture). If patient meets the osteoporosis screening criteria identified by the National Osteoporosis Foundation, they should be screened for osteoporosis with DEXA;
  * Autoimmune - patient who is currently not maintained on a medication regimen for treatment, and not stable (<6 months without exacerbation);
  * Any condition or anatomy that makes treatment with the TransLoc 3D Sacroiliac Joint Fusion System infeasible;
  * Current local or systemic infection that raises the risk of surgery;
  * Patient currently receiving disability remuneration, and/or involved in injury litigation;
  * Patient is undergoing treatment under Workman's Compensation under a claim or injury greater than 1 year;
  * Patient is participating in an investigational study or has been involved in an investigational study within 3 months prior to evaluation for participation;
  * Known to be pregnant, suspected pregnant, or planning to be pregnant prior to SIJ surgery;
  * Patient is a prisoner or a ward of the state;
  * Known or suspected drug or alcohol abuse;
  * Known allergy to titanium or titanium alloys;
  * Diagnosed psychiatric disease (e.g., schizophrenia, major depression, personality disorders) that is not well controlled for a minimum of two years and could interfere with study participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive enrollment of all patients within inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement at 12 months defined by a composite score of functional status, pain, and safety events. | 12 months
  Functional improvement and pain score have long been the standard for SI joint improvement measures. Multiple functional improvement scales will be assessed throughout the study.
Absence of Serious Adverse Events (SAEs) | From the time informed consent is signed through 12 months.
  Demonstrate safety as defined by Serious Adverse Events (SAEs).

SECONDARY OUTCOMES:
Absence of study-related adverse events | 6 months, 12 months
  Evaluate any study-related adverse events for the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Brown, DO, Principal Investigator — NY Spine and Pain Specialists
Locations (1):
- NY Spine and Pain Specialists, Port Jefferson Station, New York, United States

IPD SHARING:
Plan to Share IPD: No